CLINICAL TRIAL: NCT02950246
Title: Effect of 2% Alcoholic Chlorhexidine Compared to Povidone Iodine Solution to Limit Colonisation After Perineural Catheterization in Orthopaedic Surgery
Brief Title: Alcoholic Chlorhexidine Compared to Povidone Iodine to Limit Perineural Catheter Colonisation
Acronym: CHLOVEPI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hôpital Raymond Poincaré (Other)
Responsible Party: Principal Investigator, HARKOUK Hakim, clinical assistant chief, Hôpital Raymond Poincaré
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: CPKT-213
Record Dates: First submitted 2016-01-20; First posted 2016-11-01 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Infection of Catheter Exit Site; Catheter Related Infection
MeSH Terms: conditions — Catheter-Related Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2% alcoholic chlorhexidine group (Experimental): Skin preparation Use of 10 ml of 2% alcoholic Chlorhexidine "drug" for disinfection in place of povidone iodine without scrubing "device" Wait at least 30 secondes for drying Perineural catheterization implementation Ultrasonography use
  Interventions: Procedure: perineural catheterization implementation; Drug: 2% alcoholic chlorhexidine
- povidon iodine group (Active Comparator): Skin preparation Use of 10 ml of povidone iodine "drug" for disinfection with scrubing "device" Wait at least 30 seondes for drying Perineural catheterization implementation Ultrasonography use
  Interventions: Procedure: perineural catheterization implementation; Drug: povidon iodine

INTERVENTIONS:
Procedure: perineural catheterization implementation — Skin preparation (disinfection) with 10 ml of 2% alcoholic Chlorhexidine Perineural catheterization implementation Ultrasonography use
Drug: 2% alcoholic chlorhexidine
  Arms: 2% alcoholic chlorhexidine group
Drug: povidon iodine
  Arms: povidon iodine group

SUMMARY:
Implementation of perineural catheters may lead to infection by catheter colonization. Catheters may be colonized by the bacteria present on the skin. This is most often commensal organisms as Staphylococcus or gram negative bacilli. In a large study of 1416 peripheral nerve catheters, 28.7% of catheters were cultured positive. This colonization is most often silent because in the same study only 3% of patients had signs of local inflammation and one psoas abscess was observed (0.07%). The germs are most often coagulase negative staphylococci (61%) and gram negative bacillus (21.6%).

DETAILED DESCRIPTION:
Potential interest of alcoholic Chlorhexidine 2% to reduce the colonization of implanted catheters More recently, it is the antiseptic solution that has been the subject of several studies, including the latest on laying intravascular central catheters, highlights the superiority of alcoholic chlorhexidine 2% compared to povidone iodine alcohol [ 5]. Indeed, it was observed a reduction in the risk of bacterial infection 6 (RR 0 • 15, 95% CI 0 • 05-0 • 41) and of colonization by 5 (RR: 0.18 (95% Cl 0.13-0.24) through the use of alcoholic chlorhexidine with 2% applicator.

Such a study comparing the efficacy of the antiseptic (chlorhexidine vs Povidone-iodine) on the establishment of perineural catheters does not exist what motivated the establishment of our study.

ELIGIBILITY:
Inclusion Criteria:

* Patient classified I, II or III by the American Society of Anesthesiology
* Perineural catheterization use for pain management
* Patient should have an orthopaedic surgery

Exclusion Criteria:

* An allergy to povidone iodine
* An allergy to alcoholic Chlorhexidine 2%
* Pregnant women
* Breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-07-15 (Actual); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
perineural catheter colonization reduction | 24 months
  Assuming a frequency of the event without treatment 40%, to highlight a sub treatment relative reduction in frequency of 80% it is necessary to include 92 patients (for a 90% power and a alpha risk of 1%). According to the technique of Brun-Buisson, the catheter will be collected in a neutral tube containing 1 ml of sterile saline. In the laboratory, the tube will be vortexed for one minute and then 10μl of the sample will be seeded in oese calibrated on blood agar. Reading culture will be achieved after 48 hours at 35 ° C aerobically. The catheter will be considered settled if the count found most 1000 UFC / ml. Bacterial identification will be carried out by mass spectrometry and sensitivity by the diffusion method on Muller-Hinton agar. If there is more than one bacterial population, the number of PDUs for each bacterium was determined. In this case, we will consider only the bacterial types> 1000 UFC / ml

SECONDARY OUTCOMES:
perineural catheter infection | 24 months
  Clinical criteria of infection, redness of the puncture area or catheter insertion, hyperleukocytosis, CRP high level, fever, positive blood culture associated with positive catheter colonization, bacterial count > 1000 UFC/ml

CONTACTS AND LOCATIONS:
Overall Officials: hakim harkouk, CCA, Principal Investigator — GH Raymond Poincaré-Ambroise Paré
Locations (1):
- Chu Ambroise Pare, Boulogne-Billancourt, Île-de-France Region, France

REFERENCES:
- [Derived] Harkouk H, Thibault-Sogorb T, Beauchet A, Espinasse F, Lawrence C, Martinez V, Fletcher D. Two per cent alcoholic chlorhexidine versus alcoholic five per cent povidone-iodine for the prevention of perineural catheter colonisation: The CHLOVEPI randomised, controlled trial. Anaesth Crit Care Pain Med. 2021 Feb;40(1):100790. doi: 10.1016/j.accpm.2020.100790. Epub 2020 Dec 5. PMID 33285282